CLINICAL TRIAL: NCT04658147
Title: Feasibility and Efficacy of Perioperative Nivolumab With or Without Relatlimab for Patients With Potentially Resectable Hepatocellular Carcinoma (HCC)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J20121; IRB00246739 (Other: Johns Hopkins Medical Internal Review Board)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Relatlimab; Nivolumab; Immunotherapy; Anti PD-1; Anti - LAG-3; Resectable hepatocellular Cancer; Potentially resectable hepatocellular Cancer; Hepatocellular Cancer (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Nivolumab (Experimental): Participants receive Nivolumab only.
  Interventions: Drug: Nivolumab
- Arm B - Nivolumab and Relatlimab (Experimental): Participants receive Nivolumab and Relatlimab.
  Interventions: Drug: Nivolumab; Drug: Relatlimab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 480mg will be administered as a 30 minute IV infusion (-/+15min) at cycle 1 day 1 and at cycle 2 day 1 (28 days) then every month for up to 12 months. Intravenous administration of Nivolumab (480 mg) will occur on Cycle 1 and 2 of the study then every 28 days up to a year. Nivolumab will be administered on Day 1 of each cycle for 10 doses/ months (whichever occurs first) for adjuvant.
  Other Names: OPDIVO™; BMS 936558; MDX1106; ONO-4538
Drug: Relatlimab — Patients will receive 480 mg Relatlimab intravenously (-/+15min) on cycle 1 day 1 and at cycle 2 day 1 (every 28 days) for up to 1 year co-administered with Nivolumab.
  Other Names: BMS-986016; BMS-986016-01; Anti-LAG-3
  Arms: Arm B - Nivolumab and Relatlimab

SUMMARY:
The purpose of this study is to determine the safety and tolerability of neoadjuvant/adjuvant Nivolumab or Nivolumab plus Relatlimab in patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

• Technically resectable HCC as defined by:

* HCC may be diagnosed pathologically, or noninvasively by the American Association for the Study of Liver Diseases (AASLD) criteria or the Organ Procurement and Transplant Network (OPTN) Obligatory Diagnostic Criteria for Hepatocellular Carcinoma (HCC).

No extrahepatic spread, no nodal disease, and no bilateral left and right branch portal vein involvement.

* Measurable disease per RECIST 1.1 as determined by the investigator.
* Age ≥ 18 years old on the day of consent.
* ECOG performance status ≤1 or Karnofsky ≥80.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests prior to initial study drug.
* Patients must have adequate liver remnant and function.
* Antiviral therapy per local standard of care for hepatitis B.
* LVEF assessment with documented LVEF ≥ 50% by either TTE or MUGA (TTE preferred) within 6 months from first study drug administration.
* Woman of child-bearing potential must have a negative pregnancy test.
* Must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Fibrolamellar carcinoma or mixed HCC.
* Receiving, or previously received, any systemic chemotherapy, or investigational agent for HCC.
* Patients with a history of prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, or anti-Lag-3 antibodies.
* Has a known additional malignancy that is expected to require active treatment within two years, or is likely to be life-limiting in the opinion of the treating investigator. Superficial bladder cancer, non-melanoma skin cancers, or low grade prostate cancer not requiring therapy would not exclude participation in this trial.
* History of HIV infection.
* Active co-infection with HBV and HDV.
* Has a diagnosis of immunodeficiency, or is receiving systemic steroid therapy.
* Prior tissue or organ allograft or allogeneic bone marrow transplantation.
* History of any autoimmune disease requiring systemic treatment within the past 2 years.
* Systemic or topical corticosteroids at immunosuppressive doses (> 10 mg/day of prednisone or equivalent).
* Confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent.
* Uncontrolled intercurrent illness.•
* Uncontrolled or significant cardiovascular disease.
* Significant heart disease.
* Moderate or severe ascites.
* Known or suspected hypersensitivity to study treatment.
* Are pregnant or breastfeeding.
* WOCBP and men with female partners (WOCBP) who are not willing to use contraception.
* Unable to have blood drawn.
* Any other sound medical, psychiatric, and/or social reason as determined by the Investigator.
* Any illicit drugs or other substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who complete pre-op treatment and proceed to surgery | 4 years

SECONDARY OUTCOMES:
Number of participants experiencing study drug-related toxicities | 4 years
  Number of participants experiencing study drug-related adverse events Grade 3 or higher as defined by CTCAE v5.0.
Percentage of participants who obtain R0 resection | 8 weeks
Percentage of evaluable patients who obtain a pathologic complete response (pCR) or major pathologic response (MPR) | 8 weeks
Objective response rate (ORR) at 8 weeks | 8 weeks
  ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Overall survival (OS) at 12 months | 12 months
  OS will be measured from date of first dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Overall survival (OS) at 18 months | 18 months
  OS will be measured from date of first dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Overall survival (OS) at 3 years | 3 years
  OS will be measured from date of first dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Overall survival (OS) at 5 years | 5 years
  OS will be measured from date of first dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Disease free survival (DFS) at 12 months | 12 months
  Number of months from the date of first treatment until disease recurrence at 12 months. Estimation based on the Kaplan-Meier curve.
Disease free survival (DFS) at 18 months | 18 months
  Number of months from the date of first treatment until disease recurrence at 18 months. Estimation based on the Kaplan-Meier curve.
Disease free survival (DFS) at 3 years | 3 years
  Number of months from the date of first treatment until disease recurrence at 3 years. Estimation based on the Kaplan-Meier curve.
Disease free survival (DFS) at 5 years | 5 years
  Number of months from the date of first treatment until disease recurrence at 5 years. Estimation based on the Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yarchoan, MD, Principal Investigator — SKCCC Johns Hopkins Medical Institution
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No